CLINICAL TRIAL: NCT01769027
Title: Antibiotic Treatment and Intravenous Immunoglobulin Double-blind, Randomized, Placebo-controlled Trial for PANDAS
Brief Title: Antibiotic Treatment and Intravenous Immunoglobulin Trial for PANDAS
Acronym: ATIVPANDAS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: CNS Onlus (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Stefano Pallanti, Associate Professor, CNS Onlus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: spallanti
Record Dates: First submitted 2012-12-14; First posted 2013-01-16 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Pandas
MeSH Terms: conditions — Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections | interventions — Penicillins; Azithromycin; Sertraline; Penicillin G Benzathine; Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SSRI+AB (Active Comparator): Intervention: sertraline+antibiotic (penicillin/azithromycin) 12 weeks treatment with a combination of sertraline (to a maximum of 200 mg/day)and one antibiotic ( benzathine penicillin G 1.200.000 U every 3 weeks or, in case of allergy, azithromycin 500 mg/week ). Patients who will not respond to SSRI+antibiotic (penicillin/azithromycin) will be treated with IVIG (2g/kg over 5 days for 5 consecutive months)
  Interventions: Drug: Sertraline+Antibiotic (penicillin/azithromycin); Biological: IVIG
- SSRI+placebo (Placebo Comparator): Intervention: Sertraline+placebo 12 weeks treatment with a combination of sertraline (to a maximum of 200 mg/day) and a placebo
  Interventions: Drug: Sertraline+placebo

INTERVENTIONS:
Drug: Sertraline+Antibiotic (penicillin/azithromycin) — 12 weeks treatment with a combination of Sertraline (to a maximum of 200 mg/day) and an antibiotic (benzathine penicillin G 1.200.000 U every 3 weeks or, in case of allergy, azithromycin 500 mg/week.
  Non-responder patients will be treated with IVIG (2g/kg over 5 days for 5 consecutive months)
  Other Names: Zoloft; Lustral; Bicillin L-A; Permapen; Zythromax
  Arms: SSRI+AB
Drug: Sertraline+placebo — 12 weeks treatment with a combination of sertraline (to a maximum of 200 mg/day) and placebo
  Other Names: Zoloft; Lustral
  Arms: SSRI+placebo
Biological: IVIG — Patients who will not respond to SSRI+antibiotic (penicillin/azithromycin) will be treated with IVIG (2g/kg over 5 days for 5 consecutive months)
  Other Names: Gamimune N; Gammagard
  Arms: SSRI+AB

SUMMARY:
An increasing body of evidence indicates that an immune basis might underline a number of pediatric neuropsychiatric disorders. Research studies found a subgroup of children who had Obsessive compulsive (OCD) and/or tic disorders following a Group A beta-hemolytic streptococcal (GAS) infection. The subgroup is identified by the acronym, PANDAS (pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections. More recently, several PANDAS variants have been described, including adult-onset variant. There are many evidences that OCD/tic symptoms could be due to an immunologic reaction against brain tissues following a streptococcal infection.

The purpose of this study is to know if sertraline (one of the SSRI approved by FDA to improve OCD/tic symptoms in these patients) plus antibiotic (benzathine penicillin G or azithromycin in case of penicillin allergy) is more effective than SSRI only.

Patients who will not respond to antibiotic will be treated with intravenous immunoglobulin (IVIG) in order to inactivate the immune reaction versus brain tissues.(No treatment response is based on the lack of a Y-BOCS score improvement of at least 35%).

Objectives:

* To determine the safety and efficacy of SSRI+AB compared to SSRI only.
* To test the safety and additional beneficial effects of high dose of IVIG on antibiotic prophylaxis for the treatment of OCD symptoms in non-responders patients with PANDAS.

Study methodology:

* Participants will be screened to obtain medical history and other information at Neurologic and Psychiatric Sciences Department of Florence University Hospital and at Paris-est University.
* Participants will receive a treatment of either SSRI+AB or SSRI+placebo for 12 weeks (double-blind randomized trial)
* Patients who will not respond to AB will be admitted to the hospital to receive IVIG for 5 days, for 5 consecutive months.
* Follow-up visits will take place 3 and 6 months after the first evaluation, followed by 6 months follow-ups for 3 additional years.

Blood samples (including blood cytokine determination), ECG, Doppler and 2-dimensional echocardiogram EEG, imaging studies (2 tesla MRI), and other tests will be performed both before and after the treatment with SSRI+AB or SSRI+placebo and in case also after IVIG treatment.

DETAILED DESCRIPTION:
Inclusion criteria for PANDAS subjects are:

* Ages 4 -40 years
* Presence of DSM-IV-R obsessive compulsive disorder or tic disorder and at least two of the following:

  1. Anxieties e.g. new onset separation anxiety
  2. Sensory abnormalities (tactile/auditory/visual defensiveness or visual misperceptions)
  3. Behavioral Regression (e.g. new onset impulsivity, hyperactivity, meltdowns)
  4. Deterioration in school performance or in handwriting
  5. Emotional lability and/or depression
  6. Urinary symptoms (frequent urination or enuresis)
  7. Sleep disturbances
  8. Anorexia
* Sudden onset of symptoms or episodic course of symptom severity following infections.
* Symptoms are of moderate severity with Yale-Brown Obsessive Compulsive Scale (Y-BOCS) (or with the children's version for subjects below 16 years of age) of more or equal to 16 and/or Yale Global Tic Severity Scale (YGTSS) of more or equal to 21 and with significant impairment (CGI of moderate or worse).
* Laboratory documentation of infection as documented by at least two of these: positive throat culture, documented rise in one or more anti-GAS antibody titers such as anti-streptolysin O, anti-streptococcal DNAaseB.

Exclusion criteria for all subjects are: non-tic neurologic disorder, presence of immunologic disorder, presence of serious medical illness, IgA deficiency (< 20mg/dL), hyperviscosity syndromes, psychotropic therapy.

Interventions:

All patients will be treated with sertraline (to a maximum of 200 mg/day. This study will involve a 12 week double-blind, placebo-controlled, randomized trial with benzathine penicillin G (1.200.000 U every 3 weeks) or azithromycin (500 mg/week) in case of penicillin allergy. Non-responders patients will be treated with IVIG (2 g/kg of body weight over 5 days, for 5 consecutive months)

Outcomes:

Primary Outcome Measures:

* Significant reduction of OC/tic symptoms severity, as assessed by YBOCS/YGTSS, compared to placebo, after antibiotic prophylaxis. [ Time Frame: 6 months ]
* Significant reduction of OC/tic symptoms severity, as assessed by YBOCS/YGTSS, compared to placebo, after IVIG treatment. [ Time Frame: 6 months ]

Secondary Outcome Measures:

* The degree of treatment response is expected to correlate with the percentage reduction in antibodies titers following IVIG administration. [ Time Frame: 6 months]
* The degree of treatment response is also expected to correlate with decreased inflammation in specific regions of the brain, as demonstrated by macroscopic changes and microstructural alterations on MRI and serum and CSF cytokines and chemokines [ Time Frame: 6 months ]

Expected impact:

* To clarify the utility of antibiotic and IVIG therapy in PANDAS and how the IVIG produce their effects.
* To individualize the treatment.
* To disseminate new data for the treatment of PANDAS.

ELIGIBILITY:
Inclusion Criteria:

* Ages 4 -40 years
* Presence of DSM-IV-R obsessive compulsive disorder or tic disorder and at least two of the following:

  1. Anxieties e.g. new onset separation anxiety
  2. Sensory abnormalities (tactile/auditory/visual defensiveness or visual misperceptions)
  3. Behavioral Regression (e.g. new onset impulsivity, hyperactivity, meltdowns)
  4. Deterioration in school performance or in handwriting
  5. Emotional lability and/or depression
  6. Urinary symptoms (frequent urination or enuresis)
  7. Sleep disturbances
  8. Anorexia
* Sudden onset of symptoms or episodic course of symptom severity following infections
* Laboratory documentation of infection

Exclusion Criteria:

* Exclusion criteria for all subjects are: non-tic neurologic disorder, presence of immunologic disorder, presence of serious medical illness, IgA deficiency (< 20mg/dL), hyperviscosity syndromes, psychotropic therapy.

Ages: 4 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The improvement of OC/tic symptoms will be superior in patients treated with SSRI+AB and in case with IVIG, compared with those treated with SSRI+placebo, as assessed by the YBOCS/YGTSS | 6 months

SECONDARY OUTCOMES:
The degree of treatment response is expected to correlate with the percentage reduction in antibodies titers following IVIG administration | 6 months
The degree of treatment response is also expected to correlate with decreased inflammation in specific regions of the brain, as demonstrated by macroscopic changes and microstructural alterations on MRI and serum and CSF cytokines and chemokines | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Pallanti, MD; PhD, Principal Investigator

REFERENCES:
- [Background] Garvey MA, Perlmutter SJ, Allen AJ, Hamburger S, Lougee L, Leonard HL, Witowski ME, Dubbert B, Swedo SE. A pilot study of penicillin prophylaxis for neuropsychiatric exacerbations triggered by streptococcal infections. Biol Psychiatry. 1999 Jun 15;45(12):1564-71. doi: 10.1016/s0006-3223(99)00020-7. PMID 10376116
- [Background] Perlmutter SJ, Leitman SF, Garvey MA, Hamburger S, Feldman E, Leonard HL, Swedo SE. Therapeutic plasma exchange and intravenous immunoglobulin for obsessive-compulsive disorder and tic disorders in childhood. Lancet. 1999 Oct 2;354(9185):1153-8. doi: 10.1016/S0140-6736(98)12297-3. PMID 10513708
- [Background] Snider LA, Lougee L, Slattery M, Grant P, Swedo SE. Antibiotic prophylaxis with azithromycin or penicillin for childhood-onset neuropsychiatric disorders. Biol Psychiatry. 2005 Apr 1;57(7):788-92. doi: 10.1016/j.biopsych.2004.12.035. PMID 15820236
- [Background] Swedo SE, Leonard HL, Garvey M, Mittleman B, Allen AJ, Perlmutter S, Lougee L, Dow S, Zamkoff J, Dubbert BK. Pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections: clinical description of the first 50 cases. Am J Psychiatry. 1998 Feb;155(2):264-71. doi: 10.1176/ajp.155.2.264. PMID 9464208